CLINICAL TRIAL: NCT03031275
Title: Long-term Follow Up of Adult Patients Treated With Extracorporeal Membrane Oxygenation for Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Bernhard Holzgraefe, MD, PhD, Karolinska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2013/2258-31/1
Record Dates: First submitted 2017-01-10; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Long Term Adverse Effects; Pneumonia; Acute Respiratory Distress Syndrome; Sepsis; Critical Illness; Cognitive Impairment; Extracorporeal Circulation; Complications
Keywords: extracorporeal circulation; critical care outcomes
MeSH Terms: conditions — Long Term Adverse Effects; Pneumonia; Respiratory Distress Syndrome; Sepsis; Critical Illness; Cognitive Dysfunction | interventions — Magnetic Resonance Spectroscopy; Neuropsychological Tests

STUDY DESIGN:
Who Masked: Investigator
Masking Description: All investigators (radiologist, neuropsychologist, physiotherapist) were masked from all patient details other than the fact that they were treated with ECMO (ie did not know when the patient was treated, for what condition, if any side effects were seen and so on).

INTERVENTIONS:
Radiation: High-resolution computed tomography — HRCT of the thorax
Radiation: Magnetic resonance imaging — MRI of the brain
Behavioral: Cognitive testing — Neuropsychological testing

SUMMARY:
Follow-up after treatment with Extracorporeal Membrane Oxygenation (ECMO) at the ECMO Center Karolinska.

Patients: adult survivors treated with ECMO for severe refractory respiratory failure at least 5 years earlier.

Investigations: brain and pulmonary radiographic morphology, cognitive testing, pulmonary function testing, exercise tolerance, quality of life and mood disorder screening.

DETAILED DESCRIPTION:
All adult patients treated at the ECMO Center Karolinska between 1995 and July 2009 were screened for eligibility in January 2014. Patients living abroad (including non-Swedish citizens), patients treated for non-respiratory conditions, diseased patients and patients with a known pre-ECMO mental handicap were excluded.

Eligible patients were contacted, and patients who agreed to participate gave their written informed consent. All studied patients underwent the same study protocol during a day at the hospital, including a clinical interview, MRI scan of the brain, HRCT scan of the thorax, pulmonary function testing, neuropsychological examination, walking test, self assessment questionnaires for quality of life, anxiety, depression and post-traumatic stress.

Patient charts were reviewed for relevant clinical information, including age, gender, ECMO mode (venovenous or venoarterial), time in hospital, on ECMO, non-ECMO ICU and on mechanical ventilation; preexisting diseases, blood gas values and ventilator settings before initiation of ECMO treatment. Hand written clinical data from the patients´ charts from every hour with ECMO treatment was reviewed for ventilator settings, lung volumes, mean arterial pressure, hemoglobin, lactate and oxygenation parameters during an observation period, which was defined as the first 10 days on ECMO (or the entire treatment period if shorter than 10 days). This information was added to a digital database for the purpose of this study.

At the time of ECMO treatment, arterial hemoglobin oxygen saturation was measured by peripheral pulse oximetry from the right ear, finger or nose. Venous preoxygenator lactate and venous saturation values were used as indicators of sufficient (lactate < 2 mmol l-1 , SvO2 ≥ 70%) or insufficient tissue perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients treated with ECMO at the ECMO Center Karolinska 1995 - July 2009

Exclusion Criteria:

* Diseased patients
* Patients living abroad (including non-Swedish citizens)
* Patients treated for non-respiratory conditions
* Patients with a known pre-ECMO mental handicap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal cognitive functioning assessed by the Wechsler Adult Intelligence Scale and memory tests | 5-17 years after treatment
  Wechsler Adult Intelligence Scale, 4th ed, Rey Auditory Verbal Learning Test (learning trials 1 to 5 and delayed recall), immediate recall from the Rey Complex Figure and Logical Memory I and II from Wechsler Memory Scale, 3rd ed.
Number of participants with abnormal brain imaging assessed by magnetic resonance imaging | 5-17 years after treatment
  Sagittal and axial T1- and T2-weighted images, and coronal T2-weighted and T2-weighted fluid attenuated inversion recovery (FLAIR) images. Slice thickness 4 mm. Presence of hypoxic or anoxic damage, infarctions, hemorrhages, and contusion damage were described.
Number of Participants With Abnormal Pulmonary function | 5-17 years after treatment
  Static and dynamic spirometry. Measured results as % of the expected normal values were presented.
Number of Participants With Abnormal Lungs radiographic findings assessed by high-resolution CT scan | 5-17 years after treatment
  Non-contrast spiral scan. A series for grading of pulmonary changes was reconstructed, using a high spatial resolution reconstruction algorithm with 1 mm-width, overlapping slices. Four patterns were mapped: reticular, ground-glass opacification, consolidation and decreased attenuation.
Number of participants with signs of post-traumatic stress assessed by the Trauma Screening Questionnaire | 5-17 years after treatment
Number of participants with signs of a reduced health related quality-of-life, assessed by the Short Form-36 | 5-17 years after treatment
Number of participants with signs of a reduced Health related quality-of-life, assessed by the S:t George´s Respiratory Questionnaire | 5-17 years after treatment
Number of participants with signs of a reduced exercise tolerance | 5-17 years after treatment
  6-minute walking test
Number of participants with signs of anxiety and depression assessed by the Hospital and Anxiety Depression Scale | 5-17 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- ECMO Center Karolinska, Stockholm, Sweden